CLINICAL TRIAL: NCT05362188
Title: Efficacy and Safety of Topical Nicotinamide in Treatment of Discoid Lupus Erythematosus
Brief Title: Topical Nicotinamide in Treatment of DLE
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed Hassan Nouh MD, the principal investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 27042022
Record Dates: First submitted 2022-04-26; First posted 2022-05-05 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Discoid Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Discoid | interventions — Niacinamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Topical Nicotinamide 2% (Experimental): will receive topical nicotinamide 2%
  Interventions: Drug: Nicotinamide Topical
- Topical Nicotinamide 4% (Experimental): will receive topical nicotinamide 4%
  Interventions: Drug: Nicotinamide Topical
- Placebo (Placebo Comparator): Subjects will receive only cream/gel base without API for control
  Interventions: Drug: Nicotinamide Topical

INTERVENTIONS:
Drug: Nicotinamide Topical — Patients with discoid lupus erythematosus (face & scalp) will be given topical nicotinamide in two concentrations (2&4%) to apply twice daily for 12 consecutive weeks and then follow up.
  Topical nicotinamide will be prepared in different forms (cream & gel).
  Other Names: Topical treatment of skin lesions

SUMMARY:
Cutaneous lupus erythematosus (CLE) is lupus affecting the skin. In this autoimmune disease, the body's immune system attacks healthy skin. There are 3 main types: Acute cutaneous lupus, Subacute cutaneous lupus, and Chronic cutaneous lupus ("discoid lupus"). Lupus most often appears between the ages of 20 and 50 years; it affects women more than men, and it may happen more in patients with a family history of lupus or other autoimmune diseases.

DETAILED DESCRIPTION:
DLE is the most common form of chronic cutaneous erythematosus and can occur as a localized form (80%) with lesions on the face, ears, and scalp or as disseminated DLE (20%) with lesions above and below the neck. The disseminated form of DLE, especially when involving the trunk, is associated with an increased risk of progression to SLE. It is unusual for discoid lesions to be present below the neck without lesions also being present above the neck. Occasionally, discoid lesions develop on mucosal surfaces, including the lips, nasal mucosa, conjunctivae, and genital mucosa. Some patients with discoid lesions exhibit a photodistribution. Sun exposure seems to play a role in the development of lesions.

For discoid lupus erythematosus without associated SLE (CDLE), the evidence does not show whether circulating inflammatory cells and autoantibodies are involved in the pathogenesis, but it is evident that the cutaneous inflammatory infiltrates are dominated by Th1.

The first morphological sign of DLE is a well-defined, annular erythematous patch or plaque of varying size followed by follicular hyperkeratosis, which is adherent to the skin. By removing the adherent scale, follicle-sized keratotic spikes similar to carpet tacks can be seen ("carpet tack sign"). The lesions slowly expand with active inflammation and hyperpigmentation at the periphery leaving depressed central atrophy and scarring, telangiectasia, and hypopigmentation. DLE can progress to irreversible scarring alopecia on the scalp. Although uncommon, a squamous cell carcinoma can develop in a longstanding discoid lesion.

A biopsy from the lesion for routine histologic examination is usually diagnostic of DLE. Atrophic epidermis, keratotic plugging of the follicles, hydropic degeneration of the basal cells, and patchy perivascular and perifollicular lymphocytic infiltrate are characteristic.

Early treatment of discoid lupus lesions may lead to the total clearing of skin lesions, but treatment failure results in permanent scarring. Hair loss, depressed scars, and pigmentary changes are often disfiguring, particularly in darker-skinned people. Some general measures, such as sun avoidance and liberal application of sunscreen, are encouraged because cutaneous lesions are known to be exacerbated by sunlight. Smoking cessation is encouraged, as this can increase DLE disease activity.

While antimalarials such as hydroxychloroquine have been widely used as a first-line treatment for lupus-associated skin lesions, 30% of patients with lupus do not respond to this medication. Other available therapies such as corticosteroids and thalidomide can also be applied, however, their toxic side effects limit their clinical use. Recent studies by the investigators have shown that nicotinamide, a water-soluble vitamin whose side effects are considered minimal, can protect against skin lesions and autoantibody production. Thus it is hypothesized that nicotinamide treatment could be a novel therapy for lupus-associated skin lesions in patients with LE.

Nicotinamide is the amide form of vitamin B3 . It is the precursor of numerous reactions in the body including adenosine triphosphate (ATP) production and consequently can be used in many dermatological disorders.

ELIGIBILITY:
Inclusion Criteria:

* Age: between 18 years and 65 years old
* Patients clinically and histopathologically newly diagnosed as DLE
* Patients clinically and histopathologically diagnosed with cutaneous lupus erythematosus that has not responded to treatment with hydroxychloroquine(200-400mg/day) plus corticosteroid at a dosage less than the equivalent of (0.5mg/kg/day) for the preceding two months or a longer period

Exclusion Criteria:

* Age < 18 years old
* Pregnant and lactating women
* A history of treatments with multivitamins in the recent month
* Soft tissue infection
* Severe comorbidities including heart failure, respiratory failure
* Acute severe infections such as cellulitis or a history of HBV or HCV

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Severity index | from base line ( visit 0 ) to 1 , 2 respectively
  A change in discoid lupus erythematosus severity index
Activity score | from base line ( visit 0 ) to 1 , 2 respectively
  A change in discoid lupus erythematosus activity score

SECONDARY OUTCOMES:
Response | 2 months
  defined as > 25% change in activity score at the end of treatment
Remarkable response | 2 months
  defined as > 50% change in activity score
The dermatology life Quality Index score | 2 months
  A change in Dermatology life Quality Index score as it reflects the quality of life related to skin manifestations

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Hassan Nouh, MD, Principal Investigator — Al-Azhar university Hospital
Locations (1):
- AL-Azhar University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No